CLINICAL TRIAL: NCT04889443
Title: How do Cartilage Injuries Heal Naturally? An Observational Study of Spontaneously Healing Cartilage Defects
Brief Title: Spontaneous Healing of ARticular Cartilage (SHARC)
Acronym: SHARC
Status: Completed | Type: Observational
Sponsor: Keele University (Other)
Collaborators: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RG-0238-17-ISTM; 18/NW/0291 (Other: REC North west - Liverpool East); 243678 (Other: Health Research Authority (HRA) UK); MR/N02706X/1 (Other Grant/Funding Number: MRC UK)
Record Dates: First submitted 2021-05-07; First posted 2021-05-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Cartilage Damage; Cartilage Injury
Keywords: Cartilage repair

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cartilage repair tissue biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgical cartilage repair procedure requiring harvest procedure or Autologous Stromal Cell Implantation — Any surgical cartilage repair procedure of the knee that requires a harvest biopsy of knee cartilage, which will leave a controlled small cartilage injury
  Other Names: Autologous Chondrocyte Implantation (ACI), Matrix Assisted Chondrocyte Implantation (MACI)

SUMMARY:
SHARC is an observational study of cartilage patients who are treated with surgery that involves obtaining a harvest biopsy. SHARC will study the natural healing process of the harvest biopsy site based on histological and biochemical analyses of repair tissue biopsies, synovial fluid biomarkers, medical imaging (MRI) and gait analysis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a very common disease of the joints, for which in the United Kingdom alone almost 9 million people have sought treatment. This painful disease affects the cartilage and bone inside the joint. Many factors are known to increase the risk of getting osteoarthritis, or the rate at which it gets worse. Very important among these factors is an injury or a defect of the cartilage. It was believed for hundreds of years that cartilage, once injured, does not heal.

Research from the past 10 years is now throwing doubt on this old certainty, as researchers who took regular scans of volunteers over time noted that sometimes these defects come and then go. A Japanese group of surgeons decided to look again after a year to see what had happened to these defects, and noted that about half of them had got better! Cartilage defects in human therefore can heal, but nobody knows how this works.

For many years, our Center has helped patients who have knee cartilage damage by using the patients' own cartilage cells to help repair areas of damaged cartilage. This cell therapy starts by taking a piece of cartilage (10 mm) from the patient's knee, and this created defect always heals after a year. Thus, our proposal is to use our cell therapy patients as a human experimental model of natural cartilage healing using a wide range of techniques including Magnetic Resonance Imaging (MRI), visual inspection of the joint itself during knee joint surgery, examining biopsies of repair tissue down the microscope and measuring various kinds of molecules researchers think are important. The information gathered from these tests will help bridge the gap in our understanding of the mechanisms involved in the cartilage tissue regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Being able to provide signed and dated informed consent form.
* Scheduled for one of the following surgical treatments

  * Surgery that involves the harvest of cartilage tissue as part of the treatment, thus creating a fresh cartilage defect, which is then left to heal naturally. Examples of such surgery are autologous chondrocyte implantation (ACI) and mosaicplasty.
  * Autologous stromal cell implantation (ASCI), as part of the ASCOT randomised clinical trial.

Exclusion Criteria:

* Inadequate understanding of verbal explanations or written information given in English, or having special communication needs.
* Chronic severe renal insufficiency
* Anything that would preclude the individual's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery that involves the harvest of cartilage tissue as part of the treatment
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Fraction of hyaline cartilage in harvest repair tissue | 1 year after tissue harvest
  Fraction of hyaline or mixed hyaline/fibrous cartilage in a 1-year biopsy assessed using OsScore cartilage histology criteria

SECONDARY OUTCOMES:
Visual quality of the repair tissue in harvest repair tissue | 1 year after tissue harvest
  Visual quality of the repair tissue in a tissue biopsy obtained at 1 year, assessed using the corresponding item in the International Cartilage Repair Society (ICRS)-II arthroscopy score.
Quality of harvest repair tissue assessed from MRI images | 1 year after tissue harvest
  The quality of the repair tissue assessed from MRI images using the Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) score obtained at 1 year.
Mean signal intensity of harvest repair tissue on MRI | 1 year after tissue harvest
  The mean signal intensity of the repair tissue on an MRI T2 map obtained at 1 year
Quality of harvest repair tissue assessed from a biopsy using the ICRS-II histology score | 1 year after tissue harvest
  Quality of repair tissue assessed from a tissue biopsy at 1 year by the total ICRS-II histology score (ordinal scale from 0 to 140).
Quality of harvest repair tissue assessed from a biopsy using the OsScore histology score | 1 year after tissue harvest
  Quality of repair tissue assessed from a tissue biopsy at 1 year by the OsScore histology score (ordinal scale from 0 to 10).
Correlation of harvest repair tissue quality with baseline risk of osteoarthritis | 1 year after tissue harvest
  Correlation of total ICRS-II histology score of a repair tissue biopsy versus the baseline risk of osteoarthritis assessed using the minimal Rotterdam prediction model.
Correlation of harvest repair tissue quality with local mechanical load at the defect | 1 year after tissue harvest
  Correlation of quality of repair tissue (outcome 3) versus local mechanical load at the defect as assessed using gait analysis at baseline and 1 year.
Match of biomarker level time course to a postulated pattern of cartilage repair, namely Inflammation-Repair-Remodelling. | 1 year after tissue harvest
  Match of the time course of biomarker levels measured at baseline, 3 month and 1 year to a postulated pattern of cartilage repair, namely Inflammation-Repair-Remodelling.
Correlation between levels of inflammatory biomarkers and inflammatory activity measured on dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) at baseline and 1 year. | 1 year after tissue harvest
  Correlation between levels of inflammatory biomarkers and inflammatory activity measured on dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) at baseline and 1 year. DCE-MRI is a non-invasive imaging technique used to determine the state of inflammation in tissue and is routinely used to assess inflammation in patients with rheumatoid arthritis. The level of inflammation will be assessed as the percentage increase in signal intensity per second from the onset of signal increase until the maximum signal.
Correlation of level of levels of inflammatory activity determined in a repair tissue biopsy versus that measured on DCE-MRI. | 1 year after tissue harvest
  Correlation between grade of inflammatory biomarkers in a repair tissue biopsy at 1 year as analysed using immunohistochemistry (IHC) and level of inflammatory activity as measured on DCE-MRI. The grade of inflammation on IHC will be assessed as the mean staining intensity per cell, and the level of inflammatory activity on DCE-MRI will be assessed as described for Outcome 10, but using a region of interest encompassing only the location of the biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Herman Kuiper, PhD, Principal Investigator — Keele University
Locations (1):
- RJAH Orthopaedic Hospital NHS Foundation Trust, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
After the study end and publication of results, individual data will be available upon request to the PI. No patient identifiable information will be shared. All individual data will be link-anonymized and a minimum of 3-way anonymization of relevant data will be used to ensure that participants cannot be identified from the supplied data.
Supporting Information: Study Protocol
Time Frame: After the study end and after the study results have been published
Access Criteria: The access will adhere to Keele University's Research Data Management Policy. Briefly, a data-sharing agreement must be issued and signed by appropriate authorities before data are released or analyses are performed on behalf of the requester.
  The Data-sharing agreement will prohibit any attempt to (a) identify study participants from the released data or otherwise breach confidentiality, (b) make unapproved contact with study participants.